CLINICAL TRIAL: NCT00085631
Title: An International Multi Center Phase III Study of Chemoradiotherapy Versus Chemoradiotherapy Plus Hyperthermia for Locally Advanced Cervical Cancer
Brief Title: Cisplatin and Radiation Therapy With or Without Hyperthermia Therapy in Treating Patients With Cervical Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was closed because of slow accrual
Sponsor: Mark Dewhirst (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Northwestern University (Other)
Responsible Party: Sponsor-Investigator, Mark Dewhirst, Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00005267; DUMC-4516 (Other: Duke Legacy IRB number); CDR0000370860 (Other: National Cancer Institute)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-07

CONDITIONS: Cervical Cancer
Keywords: stage IA cervical cancer; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Diathermy; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients received cisplatin IV and concurrently underwent hyperthermia treatment over 60-90 minutes on day 1. Patients also underwent external beam radiation therapy once daily on days 1-5. Treatment repeated weekly for 5-6 weeks in the absence of disease progression or unacceptable toxicity. After completion of chemoradiotherapy and hyperthermia, patients underwent brachytherapy to the cervix for 2-3 days.
  Interventions: Drug: cisplatin; Procedure: hyperthermia treatment; Radiation: brachytherapy; Radiation: external beam radiation therapy
- Arm II (Active Comparator): Patients received cisplatin and undergo external beam radiation therapy (and brachytherapy) as in arm I.
  Interventions: Drug: cisplatin; Radiation: brachytherapy; Radiation: external beam radiation therapy

INTERVENTIONS:
Drug: cisplatin — Given IV
  Other Names: Platinol-AQ
Procedure: hyperthermia treatment — Patients undergo hyperthermia treatment over 60-90 minutes
  Arms: Arm I
Radiation: brachytherapy — Patients undergo brachytherapy for 2-3 days
Radiation: external beam radiation therapy — Patients undergo external beam radiation therapy once daily on days 1-5

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Hyperthermia therapy kills tumor cells by heating them to several degrees above body temperature. It is not yet known whether chemotherapy and radiation therapy are more effective with or without hyperthermia therapy in treating cervical cancer.

PURPOSE: This randomized phase III trial compared the safety and efficacy of cisplatin and radiation therapy, together with hyperthermia therapy versus cisplatin and radiation therapy alone in the treatment of locally advanced cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Compare local control, failure-free survival, and overall survival of patients with locally advanced carcinoma of the cervix treated with cisplatin and radiotherapy alone, versus cisplatin and radiotherapy with hyperthermia .

OUTLINE:

This is a randomized, multicenter study. Patients are stratified according to participating center, disease stage (IIB or IIIA vs IIIB or IVA) and age (< 60 years vs ≥ 60 years). Patients are randomized to 1 of 2 treatment arms.

LIMITATIONS:

There are integrity issues with the currently available data, involving international institutions, in that several pieces of information relating to patient accrual and outcomes cannot be verified. Therefore, it would be inappropriate to report outcome measures for this study. Baseline measures of age and gender are reported for the entire study cohort. Participant flow is reported by treatment arm assignment, which was available for a majority of patients in the currently available data. Adverse events are reported for the entire cohort, as some adverse events could not be classified within a particular treatment arm.

ELIGIBILITY:
Inclusion criteria:

Invasive cervical carcinoma (squamous, adeno or adenosquamous histologies, small cell histology excluded)

* age >18years
* International Federation of Gynecology and Obstetrics ((FIGO) stage IB2, IIA-IVA, FIGO stages IA, IB1 with positive pelvic lymph nodes or parametria either on imaging techniques or pathologically involved at the time of surgery.

patients undergoing surgical removal of the cervix and uterus are not eligible, parametria either on imaging techniques or pathologically involved at the time • Performance status Eastern Cooperative Oncology Group(ECOG)/World Health Organisation (WHO) 0, 1 or >/=70%respectively White Blood count (WBC) ≥ 3,000, platelets ≥ 100,000, Absolute Neutrophil Count (ANC) > 1500

• serum bilirubin ≤ 1.5 times upper limit of normal, transaminase ≤ 3 times upper limit of normal calculated creatinine clearance >60milliliters (mls)/liter ( Cockcroft) OR creatinine </= 2.0mgs% paraaortic adenopathy absent or 1.5 centimeter (cm) in greatest dimension on Computerised Tomography (CT) or Magnetic Resonance Imaging (MRI) scan;

No history of myocardial infarction in the last 6 months no symptomatic angina pectoris negative pregnancy test in patients under 50 Hemoglobin >12.0 Gd/dl or >7.5 mmo;/L with transfusion if needed written written informed consent

Exclusion criteria:

surgical resection of the primary tumor (i.e. Total abdominal hysterectomy (TAH)/ Bilateral salpingoophorectomy (BSO)

* patients with pacemakers or implanted defibrillators
* patients with significant metallic foreign bodies (i.e. hip replacements, bone metallic rods,orthopedic plates, etc.)
* prior radiotherapy or chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2003-03; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen L. Jones, MD, PhD, Principal Investigator — Duke Cancer Institute; Leonard R. Prosnitz, MD, Principal Investigator — Duke Cancer Institute; Mark Dewhirst, DVM PhD, Principal Investigator — Duke Cancer Institute; Zeljko Vujaskovic, MD PhD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 2003 and 2008 from seven different university hospitals and medical centers internationally. A total of 101 patients were enrolled from these institutions and randomized by institution, disease stage and age.
Pre-assignment Details: Participant flow includes patients who were enrolled and randomized into the study. A third group of patients (Unavailable) was added in this participant flow to account for patients who were randomized, but whose treatment assignment was not documented in the current data.
Groups:
- Unavailable: Unavailable refers to patients who were randomized into one of the two treatment groups, but whose assignment could not be deduced from the current data. "Completed" patients were those who had documented response or follow-up data in the current dataset.
- Chemoradiation: Patients in this arm were randomized to receive cisplatin chemotherapy and radiation therapy, without hyperthermia therapy. "Completed" patients were those who had documented response or follow-up data in the current dataset.
- Chemoradiation + Hyperthermia: Patients in this arm were randomized to receive cisplatin chemotherapy and radiation therapy, together with hyperthermia therapy. "Completed" patients were those who had documented response or follow-up data in the current dataset.
Period: Overall Study
Arm/Group | Unavailable | Chemoradiation | Chemoradiation + Hyperthermia
Started | 13 | 49 | 39
Completed | 9 | 38 | 32
Not Completed | 4 | 11 | 7
Not completed — Missing Data | 4 | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Due to integrity issues with the current data, baseline measurements of age and gender are reported for the entire cohort, rather than by treatment arm. Age and gender information were available in the current documentation for all 101 patients in this study.
Arm/Group | Overall Study
Number analyzed (Participants) | 101
Age Continuous [Mean (Standard Deviation); unit: years] | 50.25 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Tumor Response Rate at 4-6 Weeks Post Treatment
Description: Primary tumor response rate is the proportion of subjects achieving a best response of complete (CR) or partial (PR) responses, according to the RECIST criteria for change in sum of longest diameters.
Time Frame: 3 months from start of therapy
Groups:
- Overall Study: Due to integrity issues with the current documented data, results are not reported for the primary tumor response rate in this study.
Arm/Group | Overall Study
Number analyzed (Participants) | 0

2. Primary Outcome: Five-year Failure-free Survival
Description: Five-year failure free survival (FFS) time was defined as the time from randomization until relapse/disease progression (local and/or distant) or death from any cause. Progression was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. The 5-year FFS rate is a percentage representing the fraction of randomized patients who, after 5 years, are disease free or alive.
Time Frame: 5 Years
Groups:
- Overall Study: Due to integrity issues with the current documented data, results are not reported for the 5-year failure-free survival rate in this study.
Arm/Group | Overall Study
Number analyzed (Participants) | 0

3. Primary Outcome: Five-Year Local Recurrence-Free Survival
Description: Five-year local recurrence-free survival (LRFS) time was defined as the time from randomization until local progressive disease or death from any cause. Local recurrence was defined as evidence of disease progression on physical exam or radiologic study, confirmed histologically by tissue biopsy. Progression was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. The 5-year LRFS rate is a percentage representing the fraction of randomized patients who, after 5 years, do not have local progression or are alive.
Time Frame: 5 years
Groups:
- Overall Study: Due to integrity issues with the current documented data, results are not reported for the 5-year local recurrence-free survival rate in this study.
Arm/Group | Overall Study
Number analyzed (Participants) | 0

4. Primary Outcome: Five-Year Overall Survival
Description: Five-year overall survival (OS) time was time from date of randomization until death from any cause. The 5-year OS rate is a percentage, representing the fraction of randomized patients who, after 5 years, are still alive.
Time Frame: 5 Years
Groups:
- Overall Study: Due to integrity issues with the current documented data, results are not reported for the 5-year overall survival rate in this study.
Arm/Group | Overall Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse events of all toxicity grades are reported for the entire cohort, as some adverse events could not be classified within a particular treatment arm.
Groups:
- Overall Study: Patients from both arms were combined in adverse event reporting.
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 10/101
Other Adverse Events (participants affected / at risk) | 54/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (N=101)
Myocardial infarction (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Allergic reaction (Immune system disorders) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Thromboembolic event (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (N=101)
"Cardiac disorders - Other, specify: Valvular heart disease" (Cardiac disorders) | 1
Blurred vision (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 15
Diarrhea (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 9
Pain (General disorders) | 7
Allergic reaction (Immune system disorders) | 1
Bronchial infection (Infections and infestations) | 1
"Infections and infestations - Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Cervix" (Infections and infestations) | 1
"Infections and infestations - Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Vulva" (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Burn (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 2
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
Weight gain (Investigations) | 1
Weight loss (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Headache (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 4
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 2
Vaginal discharge (Reproductive system and breast disorders) | 3
Vaginal hemorrhage (Reproductive system and breast disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
"Skin and subcutaneous tissue disorders - Other, specify" (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 4
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
There are integrity issues with the currently available data, involving international institutions, in that several pieces of information relating to patient accrual and outcomes cannot be verified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No